CLINICAL TRIAL: NCT06269380
Title: Evaluation of Antral Biopsies Obtained in Normal Esophagogastroduodenoscopy: A Retrospective Cohort Study
Brief Title: Evaluation of Antral Biopsies Obtained in Normal Esophagogastroduodenoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Burak Dincer, Principal investigator, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 30.01.2024-4274
Record Dates: First submitted 2024-02-12; First posted 2024-02-21 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Gastritis H Pylori; Gastritis Chronic; Intestinal Metaplasia
Keywords: Esophagogastroduodenoscopy; Routine biopsy; Intestinal metaplasia
MeSH Terms: interventions — Endoscopy, Digestive System

STUDY DESIGN:
Intervention Model Description: The biopsies obtained from patients who underwent esophagogastroduodenoscopy and were found to have normal endoscopic findings will be evaluated. The histopathological findings and their frequencies in these biopsies will be examined to assess the necessity of routine biopsy during esophagogastroduodenoscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normal esophagogastroduodenoscopy (Experimental): Patients with normal esophagogastroduodenoscopic findings and biopsy samples were obtained.
  Interventions: Procedure: Esophagogastroduodenoscopy; Procedure: Endoscopic biopsy sampling

INTERVENTIONS:
Procedure: Esophagogastroduodenoscopy — During the procedure, endoscopic examination of the upper gastrointestinal tract was made. Biopsy sampling can be made during procedure if endoscopist deemed necessary.
Procedure: Endoscopic biopsy sampling — The obtaining of biopsy samples for control purposes despite the absence of endoscopic pathology during esophagogastroduodenoscopy.

SUMMARY:
Esophagogastroduodenoscopy (EGD) is commonly performed in patients presenting with abdominal pain and dyspeptic symptoms, serving as a valuable diagnostic and therapeutic tool. While various methods are available for biopsy sampling when mucosal pathology is observed during EGD, the practice of obtaining biopsies from endoscopically normal mucosa remains controversial. Although there is literature suggesting that routine biopsies from the antrum and duodenum for surveillance purposes increase costs, pathological findings can sometimes be detected in areas that appear normal on mucosal examination, leading to potential changes in treatment approach if biopsies are obtained.

In this study, a retrospective evaluation of the prevalence of various pathologies detected in biopsies obtained from endoscopically normal mucosa in patients who underwent EGD was reported as normal.

DETAILED DESCRIPTION:
Esophagogastroduodenoscopy (EGD) is a commonly used diagnostic tool in upper gastrointestinal system diseases. Its widespread use is facilitated by its minimally invasive nature, the possibility of therapeutic procedures, low complication rates, and broad applicability. Although there are numerous guidelines regarding approaches to endoscopic pathologies and diseases detected during esophagogastroduodenoscopy, the necessity of biopsy sampling from mucosal areas that are endoscopically normal remains controversial.

In this study, patients aged between 18 and 95 who underwent EGD at the Sisli Hamidiye Etfal Training and Research Hospital Surgical Endoscopy Unit between 2021 and 2023, with no pathology detected during the endoscopic examination and who underwent biopsy sampling, will be evaluated. History of upper gastrointestinal surgery, detection of the endoscopic pathology, and not having biopsy sampling will be considered as exclusion criteria. The rate of detection of histopathological findings in the obtained biopsies, severity and activity of gastritis, rate and density of Helicobacter pylori detection, and rate and extent of intestinal metaplasia will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-95
* Endoscopically normal esophagogastroduodenoscopy
* Sampling biopsies must be obtained

Exclusion Criteria:

* History of upper gastrointestinal surgery
* Abnormal endoscopic findings such as gastritis, ulcer, hiatal hernia, pyloric deformity, alkaline reflux
* Not having biopsy

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Rate of abnormal histopathologic findings | 2 week after esophagogastroduodenoscopy
  Rate of abnormal histopathologic findings in patients with normal esophagogastroduodenoscopy and sampling biopsies obtained

SECONDARY OUTCOMES:
Rate of intestinal metaplasia | 2 week after esophagogastroduodenoscopy
  Rate of intestinal metaplasia in patients with normal esophagogastroduodenoscopy and sampling biopsies obtained
Rates of gastritis severity and activity | 2 week after esophagogastroduodenoscopy
  Rate of gastritis severity and activity in patients with normal esophagogastroduodenoscopy and sampling biopsies obtained
Rate of Helicobacter Pylori positivity | 2 week after esophagogastroduodenoscopy
  Rate of Helicobacter Pylori positivity in patients with normal esophagogastroduodenoscopy and sampling biopsies obtained

CONTACTS AND LOCATIONS:
Overall Officials: Burak Dincer, M.D., Principal Investigator — Sisli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Sisli Hamidiye Etfal Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dincer B, Omeroglu S, Guven O, Yanar C, Demir U, Akgun IE. Evaluation of Antral Biopsies Obtained in Endoscopically Normal Esophagogastroduodenoscopy: A Retrospective Cohort Study. Surg Laparosc Endosc Percutan Tech. 2024 Aug 1;34(4):439-443. doi: 10.1097/SLE.0000000000001302. PMID 38957011